CLINICAL TRIAL: NCT06545643
Title: Personalized Risk Assessment of Seizures Sensitive to Poor Sleep: a Longitudinal Study Using Wearable Electroencephalography Devices
Brief Title: Sleep-Sensitive Seizure Risk Assessment With Wearable EEGs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00115560
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy Intractable
Keywords: epilepsy; sleep; wearable EEG
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Intervention Model Description: All participants will initially undergo a screening night at a sleep lab before being equipped with a Dreem EEG headband and a Fitbit for continuous monitoring of sleep patterns and epileptic activity at home. Over 21 days, participants will wear the Fitbit daily and the Dreem headband exclusively at night as part of the data collection protocol. Additionally, participants will maintain daily sleep and seizure diaries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dreem headband (Experimental): Participants will wear a Fitbit daily and a Dreem headband exclusively at night in their homes over a 21-day period as part of the data collection protocol. Additionally, they will maintain daily sleep and seizure diaries.
  Interventions: Device: Dreem headband

INTERVENTIONS:
Device: Dreem headband — The Dreem headband is an EEG-based wearable tool that can be used to reliably assess the relationship between sleep and epilepsy over extended observation periods.

SUMMARY:
Epilepsy, a prevalent neurological disorder, affects 40% of patients with uncontrolled seizures despite medications. Sleep disturbance exacerbates epilepsy, and vice versa, but existing literature suffers from limitations. Studies conducted in hospital settings provide only brief observation periods and fail to capture the natural sleep environment. Wearable technology offers a promising solution, providing a nuanced understanding of the relationship between seizures and sleep. The Dreem headband, an EEG-based wearable, is well-suited for such studies, offering ease of use and validated accuracy. This technology enables extended observation periods under stable medication conditions, essential for assessing the complex interplay between sleep and epilepsy. By elucidating the impact of sleep on seizures, the researchers seek to identify patient populations where sleep significantly influences seizure susceptibility, ultimately informing personalized epilepsy treatments.

DETAILED DESCRIPTION:
The first aim of this study is to investigate how variations in sleep timing, duration, and structure influence seizure risk, particularly in individuals with sleep-sensitive seizures. The investigators will conduct longitudinal EEG assessments to analyze how changes in sleep features correlate with interictal epileptiform discharge rates and seizure occurrences over time.

The second aim is to develop a sleep quality index that predicts individual risk for sleep-sensitive seizures, the Sleep-Sensitive Epilepsy Risk Index (SERI). This index aims to predict an individual's seizure risk associated with disrupted sleep, facilitating personalized and preventative patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* At least 2 seizures per week based on clinical notes
* Patients where medications will stay stable over the study period
* 40% of both spikes and spindles are identifiable on the dreem headband based on the screening night

Exclusion Criteria:

* Cognitive impairment
* Psychiatric comorbidities which may influence sleep
* No bedpartner/caregiver to observe seizures
* Low agreement (below 60%) between Dreem's sleep scoring and manual scoring will be excluded from the study
* Apnea-hypopnea index of > 10/h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Total sleep time (sleep macrostructure) | 21 days
  Total sleep time as measured by the Dreem headband
Spike rates per hour (epilepsy marker) | 21 days
  Spikes will be detected by the Dreem headband
Seizure frequency per night (epilepsy marker) | 21 days
  Seizures will be detected by the Dreem headband

SECONDARY OUTCOMES:
Sleep latency (sleep macrostructure) | 21 days
  Sleep latency as measured by the Dreem headband
Wake after sleep onset (sleep macrostructure) | 21 days
  Wake after sleep onset as measured by the Dreem headband
Sleep efficiency (sleep macrostructure) | 21 days
  Sleep efficiency as measured by the Dreem headband
Sleep stage distribution (sleep macrostructure) | 21 days
  Sleep stage distribution as measured by the Dreem headband
Sleep spindle events (sleep microstructure) | 21 days
  Sleep spindles (10-16 Hz; duration 0.5-3 sec) as measured by the Dreem headband
Sleep slow wave events (sleep microstructure) | 21 days
  Slow waves (0.5-4 Hz) as measured by the Dreem headband
Performance the SERI model, as measured by the area under the receiver operating characteristic curve | Up to 2 years after study commencement
  The Sleep-Sensitive Epilepsy Risk Index (SERI) aims to predict an individual's seizure risk associated with disrupted sleep. A high SERI will indicate a high risk for sleep-sensitive seizures, while a low value will indicate a low risk.
Sensitivity of the SERI model | Up to 2 years after study commencement
  The Sleep-Sensitive Epilepsy Risk Index (SERI) aims to predict an individual's seizure risk associated with disrupted sleep. A high SERI will indicate a high risk for sleep-sensitive seizures, while a low value will indicate a low risk.
Specificity of the SERI model | Up to 2 years after study commencement
  The Sleep-Sensitive Epilepsy Risk Index (SERI) aims to predict an individual's seizure risk associated with disrupted sleep. A high SERI will indicate a high risk for sleep-sensitive seizures, while a low value will indicate a low risk.
Performance the SERI model, as measured by F1-score | Up to 2 years after study commencement
  The Sleep-Sensitive Epilepsy Risk Index (SERI) aims to predict an individual's seizure risk associated with disrupted sleep. A high SERI will indicate a high risk for sleep-sensitive seizures, while a low value will indicate a low risk.
  The F1 score ranges from 0 to 1. A value of 0 indicates poor performance, and a value of 1 represents perfect performance.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Frauscher, MD PD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No